CLINICAL TRIAL: NCT06809140
Title: Phase 2 Trial of Enfortumab Vedotin Plus Pembrolizumab With Selective Bladder Sparing for Treatment of Muscle-invasive Urothelial Cancer of the Bladder
Brief Title: Enfortumab Vedotin Plus Pembrolizumab With Selective Bladder Sparing for Treatment of Muscle-invasive Bladder Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Matthew Galsky (Other)
Collaborators: Seagen Inc. (Industry); Astellas Pharma Inc (Industry); Merck Sharp & Dohme LLC (Industry); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor-Investigator, Matthew Galsky, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCRN-GU22-598
Record Dates: First submitted 2025-01-17; First posted 2025-02-05 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Muscle Invasive Bladder Urothelial Carcinoma
Keywords: MIBC; Pembrolizumab; Enfortumab vedotin
MeSH Terms: interventions — enfortumab vedotin; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Patients with MIBC will receive 3 cycles (C1-C3) of induction enfortumab vedotin plus pembrolizumab followed by restaging including MRI of the bladder, urine cytology, and cystoscopy with TURBT of any visible tumor and/or resection site plus random biopsies using a recommended template. Patients achieving a stringently defined cCR will receive 14 cycles of "maintenance" treatment. Enfortumab vedotin will be administered during the first 6 cycles (C4-C9) of "maintenance" treatment and pembrolizumab will be given all 14 cycles (C4-C14). Patients with any residual disease at clinical restaging (i.e., >cTa disease) will undergo cystectomy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Enfortumab vedotin plus pembrolizumab (Experimental): Patients with MIBC will receive 3 cycles (C1-C3) of induction enfortumab vedotin (1.25 mg/kg for a maximum dose of 125 mg) plus pembrolizumab (200 mg) followed by restaging including MRI of the bladder, urine cytology, and cystoscopy with TURBT of any visible tumor and/or resection site plus random biopsies using a recommended template. Patients achieving a stringently defined cCR (defined below) will receive 14 cycles of "maintenance" treatment. Enfortumab vedotin (1.25 mg/kg for a maximum dose of 125 mg) will be administered during the first 6 cycles (C4-C9) of "maintenance" treatment and pembrolizumab (200 mg) will be given all 14 cycles (C4-C14). Patients with any residual disease at clinical restaging (i.e., >cTa disease) will undergo cystectomy.
  Interventions: Drug: Enfortumab vedotin; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Enfortumab vedotin — 1.25 mg/kg (maximum dose 125 mg)
Drug: Pembrolizumab — 200 mg

SUMMARY:
Patients with MIBC will receive 3 cycles (C1-C3) of induction enfortumab vedotin plus pembrolizumab followed by restaging including MRI of the bladder, urine cytology, and cystoscopy with TURBT of any visible tumor and/or resection site plus random biopsies using a recommended template. Patients achieving a stringently defined cCR (clinical complete response) will receive 14 cycles of "maintenance" treatment. Enfortumab vedotin will be administered during the first 6 cycles (C4-C9) of "maintenance" treatment and pembrolizumab will be given all 14 cycles (C4-C14). Patients with any residual disease at clinical restaging (i.e., >cTa disease) will undergo cystectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
2. Age ≥ 18 years at the time of consent.
3. ECOG Performance Status of 0-1 within 28 days prior to registration.
4. Histological evidence of clinically localized muscle-invasive urothelial cancer of the bladder clinical stage T2-3N0M0. Participants with mixed histology are eligible provided the urothelial component is ≥50% with the following exceptions: (a) tumors with any degree of squamous differentiation are eligible provided there is a urothelial cancer component, (b) tumors that contain any component of neuroendocrine histology are not eligible. N0 will be considered as the absence of radiographically enlarged lymph nodes on baseline imaging (i.e., Patients with lymph nodes ≥1 cm in short axis on imaging are not eligible).
5. Have undergone a standard of care maximal transurethral resection of bladder tumor ≤ 90 days prior C1D1. A maximal TURBT should be performed when feasible and is defined as a macroscopically complete resection of bladder tumor.
6. All subjects must have adequate transurethral resection of bladder tumor tissue available for submission identified during screening. The specimen must include tumor tissue (i.e., if a restaging maximal TURBT was performed and there was no cancer in the specimen, tissue from the most recent prior TURBT that established the diagnosis of muscle-invasive urothelial cancer of the bladder should be submitted). Tissue from both the restaging TURBT and the prior diagnostic TURBT may be requested. Subjects without available archival tissue must be discussed with the sponsor-investigator.
7. Be deemed eligible to undergo radical cystectomy and pelvic lymph node dissection
8. Demonstrate adequate organ function as defined below. All screening labs to be obtained within 28 days prior to registration.

   * Absolute neutrophil count (ANC): ≥ 1.5 x 10^9/L
   * Hemoglobin (Hgb): ≥ 9 g/dL
   * Platelets: ≥ 100 x 10^9/L
   * Creatinine clearance: ≥ 30 mL/min
   * Bilirubin: ≤ 1.5 ×ULN OR direct bilirubin ≤ ULN for participants with total bilirubin levels > 1.5 × ULN
   * Aspartate aminotransferase (AST): ≤ 2.5 × ULN
   * Alanine aminotransferase (ALT): ≤ 2.5 × ULN
   * International normalized ratio (INR) or Prothrombin time (PT) or Partial thromboplastin time (PTT): ≤ 1.5 ×ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range for intended use of anticoagulants

10. Females of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to registration. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. WOCBP must agree to use contraception.

11. Male participants able to father a child who are sexually active with female of childbearing potential must be willing to use an effective method(s) of contraception.

Exclusion Criteria:

1. Pre-existing sensory or motor neuropathy Grade ≥ 2
2. Ongoing clinically significant toxicity (Grade 2 or higher with the exception of alopecia) associated with prior treatment (including systemic therapy, radiotherapy or surgery).
3. Prior systemic chemotherapy for muscle-invasive urothelial cancer of the bladder.
4. Prior malignancy active within the previous 2 years except for locally curable cancers that have been apparently cured. Patients with intermediate or lower risk prostate cancer as defined by the National Comprehensive Cancer Network (NCCN) risk stratification guidelines may be eligible for enrollment.
5. Prior radiation therapy for bladder cancer.
6. Hemoglobin A1c ≥ 8% or hemoglobin A1c 7%-<8% with associated diabetes symptoms (polyuria or polydipsia) that are not otherwise explained
7. Active infection requiring systemic therapy.
8. Known active Hepatitis B or C infection. NOTE: Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
9. HIV-infected patients on effective anti-retroviral therapy with an undetectable viral load are eligible.
10. Has a known history of active TB (Bacillus Tuberculosis).
11. Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
12. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
13. Has received a live or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines is allowed.
14. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
15. Has severe hypersensitivity (≥ Grade 3) to pembrolizumab or enfortumab vedotin and/or any of their excipients.
16. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
17. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
18. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
19. Has had an allogenic tissue/solid organ transplant.
20. Is currently receiving an investigational agent or has received an investigational agent or used an investigational device within 28 days of study registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Complete response rate with enfortumab vedotin plus pembrolizumab for MIBC | 9 weeks
  Clinical complete response rate will be defined as cT0 or cTa (low grade) disease at the time of restaging after 3 cycles of induction enfortumab vedotin plus pembrolizumab

SECONDARY OUTCOMES:
Safety of enfortumab vedotin plus pembrolizumab | 2 years
  Safety will be determined according to the NCI Common Terminology Criteria for Adverse Events (NCI CTCAE) v5
Positive predictive value (PPV) of cCR Patients | 2 years
  Estimate the positive predictive value (PPV) of cCR for 2-year bladder-intact event-free survival
Positive predictive value (PPV) of cCR Patients | 2 years
  Estimate the positive predictive value (PPV) of cCR for 2-year metastasis-free survival
Local recurrence-free survival | 4 years
  Estimate invasive local recurrence-free survival in patients achieving a clinical complete response and forgoing immediate cystectomy. Local recurrence free survival is defined as the time from initiation of treatment until the development of invasive local recurrences in the intact bladder.
Association between clinical complete response (cCR) and bladder-intact event-free survival | 4 years
  Estimate association between clinical complete response defined as cT0 or cTa (low grade) disease at the time of restaging after 3 cycles of induction enfortumab vedotin plus pembrolizumab and bladder-intact event-free survival defined from initiation of treatment until radical cystectomy, evidence of unresectable or metastatic disease, or death due to any cause based on the Kaplan-Meier method .
Association between clinical complete response (cCR) and recurrence-free survival | 4 years
  Estimate association between clinical complete response defined as cT0 or cTa (low grade) disease at the time of restaging after 3 cycles of induction enfortumab vedotin plus pembrolizumab and recurrence free survival defined as the time from initiation of treatment until the development of invasive local recurrences in the intact bladder based on the Kaplan-Meier method.
Association between clinical complete response (cCR) and metastasis-free survival | 4 years
  Estimate association between clinical complete response defined as cT0 or cTa (low grade) disease at the time of restaging after 3 cycles of induction enfortumab vedotin plus pembrolizumab and metastasis-free survival defined as the time from initiation of treatment to the development of metastatic disease based on the Kaplan-Meier method.
Association between clinical complete response (cCR) and overall survival | 4 years
  Estimate association between clinical complete response defined as cT0 or cTa (low grade) disease at the time of restaging after 3 cycles of induction enfortumab vedotin plus pembrolizumab and overall survival defined as the time from initiation of treatment to date of death from any cause based on the Kaplan-Meier method.
Bladder-intact event-free survival | 4 years
  Bladder-intact event-free survival is defined from initiation of treatment until radical cystectomy, evidence of unresectable or metastatic disease, or death due to any cause. Bladder-intact event-free survival will be estimated in patients achieving a clinical complete response.
Pathologic stage | 4 years
  Pathologic stage will be defined based on TNM staging of the cystectomy specimen. Pathologic stage will be explained in patients who did not achieve a clinical complete response and in patients achieving a clinical complete response who subsequently undergo cystectomy.
Metastasis-free survival | 4 years
  Metastasis-free survival is defined as the time from initiation of treatment to the development of metastatic disease. Microscopic metastatic disease involving regional lymph nodes resected at cystectomy performed with curative intent will not be considered an event. Metastasis-free survival will be estimated in patients achieving a clinical complete response, in patients not achieving a clinical complete response, and in the overall cohort.
Overall survival | 4 years
  Overall survival is defined as the time from initiation of treatment to date of death from any cause. Overall survival will be estimated in patients achieving a clinical complete response, in patients not achieving a clinical complete response, and in the overall cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Galsky, MD, Principal Investigator — Sponsor-Investigator
Locations (4):
- United States (4):
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No